CLINICAL TRIAL: NCT02825147
Title: Pegaspargase and Methotrexate Based Regimens for Newly Diagnosed Extranodal NK/T Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shanghai Ruijin Hospital
Record Dates: First submitted 2015-11-22; First posted 2016-07-07 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Nasal Type Extranodal NK/T-Cell Lymphoma
Keywords: pegaspargase,methotrexate
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — pegaspargase; Methotrexate; Dexamethasone; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MESA (Experimental): stage I/II: methotrexate 1000mg/m2,d1 dexamethasone 40mg,d2-d4 etoposide 100mg,d2-d4 pegaspargase 2500U/m2,d5 a cycle of every 21 days with totally 4 cycles Radiotherapy at least 50Gy in dose for the involved local focus is sandwiched after 2 cycles.
  Interventions: Drug: Pegaspargase; Drug: Methotrexate; Drug: Dexamethasone; Drug: Etoposide; Radiation: radiotherapy

INTERVENTIONS:
Drug: Pegaspargase
Drug: Methotrexate
Drug: Dexamethasone
Drug: Etoposide
Radiation: radiotherapy

SUMMARY:
Extranodal NK/T cell lymphoma is an aggressive tumor with higher incidence in Asia.Traditional CHOP/CHOP-like regiment can't produce satisfied outcome for the patients. Asparaginase-based treatment has been demonstrated as promising response rate and survival superiority. Stage-specified regimen may bring out exciting efficacy with good safety.

DETAILED DESCRIPTION:
Extranodal NK/T cell lymphoma is a kind of tumor more prevalent in Asia and South America than that in the Western world, which is almost invariably EBV- associated and often presents as localized disease in and around the nasal structures. The disease frequency was higher in Asian countries with no differences in age, gender or immunophenotypic profile between nasal and extranasal cases. EBV is a constant finding, particularly in the cases presenting as localized nasal disease and assumed involved in the pathogenesis. During the past decades the disease, historically termed as "lethal midline granuloma" was very aggressive with poor survival. Five-year OS for extra-nasal disease is reported as 9% compared to 42% for localized disease.

Although radiotherapy combined with or without anthracycline-based chemotherapy has been considered as the treatment for extranodal NK/T cell lymphoma in the past, numerous data suggest that this tumor is not very chemosensitive due to the p-glycoprotein expression, which may mediate the drug resistance. CHOP/CHOP-like schedules presented with low CR rates and frequent failures during chemotherapy. Disseminated involvement is much poorer in prognosis than localized disease with the latter is benefit more from radiotherapy.

In the nearest ten years, many new agents have been used in the treatment of extranodal NK/T cell lymphoma, in which the most promising one is asparaginase. Asparaginase-containing regiment has demonstrated about 50% responses rates and 5-year overall survival of 65% in relapsed or refractory disease. The impressive outcome indicates its value in the newly diagnosed patients, especially in the disseminated cases. Pegaspargase as a new form of asparaginase displays equivalent bioactivity as L- asparaginase with longer half-time and lower incidence of allergy. Its clinical efficacy has been verified in the patients with acute lymphocytic leukemia.

The purpose of this study is to evaluate the efficacy and safety of pegaspargase and methotrexate based regimens with or without radiotherapy in the newly diagnosed patients with extranodal NK/T cell lymphoma, including localized and disseminated cases.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of extranodal NK/T cell lymphoma, nasal type, previously untreated
* Age 14 ~ 70 years old
* ECOG(Eastern Cooperative Oncology Group）performance status 0~2
* Stage I to II
* Life expectancy>6 months
* Informed consented

Exclusion Criteria:

* Chemotherapy before
* Bone marrow transplantation before
* History of malignancy
* Uncontrollable cardio-cerebral vascular, coagulative, autoimmune, serious infectious disease
* LVEF≤50%
* Other uncontrollable medical condition that may that may interfere the participation of the study
* Lab at enrollment ALT or AST >3*ULN, AKP or bilirubin >2.5*ULN Creatinine>1.5*ULN
* Not able to comply to the protocol for mental or other unknown reasons
* Pregnant or lactation
* HIV infection

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 21 days after 4 cycles of chemotherapy

SECONDARY OUTCOMES:
Progression free survival | 2-year
overall survival | 2-year
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Day 1 of each course and then every 3 months for 1 years

CONTACTS AND LOCATIONS:
Overall Officials: ZHAO WEILI, PhD,MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, China